CLINICAL TRIAL: NCT06471816
Title: Promoting Mental Health in Young Children - a Dialogue Based Approach in Kindergartens: A Randomized Controlled Trial
Brief Title: Promoting Mental Health in Young Children - a Dialogue Based Approach in Kindergartens
Acronym: PRO-DIALOG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Collaborators: University of Bergen (Other); Western Norway University of Applied Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 151749
Record Dates: First submitted 2024-06-18; First posted 2024-06-24 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Child Behavior; Child Development
Keywords: Health Promotion; Secondary Prevention; Kindergarten; Child Mental Health; Parent Involvement
MeSH Terms: conditions — Child Behavior

STUDY DESIGN:
Intervention Model Description: Kindergartens from three different organisations are involved. The kindergartens are randomized to the implementation or control condition within each organisation (block randomization).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention kindergartens (Experimental): Participants (parents of kindergarten children) will take part in the biannual DBED parent-teacher meetings.
  Interventions: Other: Dialogue Based Early Detection
- Control kindergartens (Active Comparator): Participants (parents of kindergarten children) will take part in traditional parent-teacher meetings.
  Interventions: Other: Traditional parent-teacher meeting

INTERVENTIONS:
Other: Dialogue Based Early Detection — Before the biannual parent-teacher meeting, both the kindergarten teacher and the parents will complete the Early Worry Questionnaire containing 39 items related to development and well-being of the individual child. For each item the respondents are asked to indicate if they during the last three months have been concerned. In the parent-teacher meeting they will discuss their possible concerns and try to reach an agreement on how to evaluate the child. If necessary, possible supportive interventions or further assessments locally in the kindergarten or in the public services will be decided.
  Arms: Intervention kindergartens
Other: Traditional parent-teacher meeting — This is an annual or biannual meeting that is prepared by the kindergarten teacher where (s)he reports on the child's appearance / behaviour and possible challenges as to development and behaviour from an educationalist's view. There are no common templates for the agenda of such meetings, however, usually the kindergarten teacher's perspective and opinion will dominate.
  Arms: Control kindergartens

SUMMARY:
The goal of this clinical trial is to learn if the novel Dialogue Based Early Detection (DBED) method can prevent impaired mental health in kindergarten children. It will also learn about the screening properties of DBED to identify children with impaired mental health, if DBED facilitates early interventions, and if DBED is well accepted and sustainable in an ordinary kindergarten setting.

The main questions it aims to answer are:

* Do children in kindergartens where DBED is implemented develop better mental health scores than children in kindergarten where DBED is not implemented?
* How well identifies DBED kindergarten children with impaired mental health compared to a traditional screening instrument (the Strengths and Difficulties Questionnaire)?
* What is the impact of DBED on activation of interventions for mental health problems?
* What is the social validity of DBED?

Researchers will compare outcomes in kindergartens where DBED is implemented with outcomes in kindergartens where it's not.

* During the last three years of kindergarten attendance participants (parents of kindergarten children) in the intervention kindergartens will take part in the biannual DBED parent-teacher meetings, while participants in the control kindergartens will take part in traditional parent-teacher meetings.
* Twice a year all participants will answer questionnaires of the child's mental health and parental stress during the follow-up period (3 years in kindergarten and 2 first years in school).
* Participants in the intervention kindergartens will answer user satisfaction questionnaires after every parent-teacher meeting.
* The kindergarten teachers will report on type and time of supportive interventions for each participating child during the follow-up period in kindergarten.

ELIGIBILITY:
Inclusion Criteria:

* Attendance in kindergarten
* Inclusion during the first half-year of the third last year in kindergarten

Exclusion Criteria:

* Parents don't communicate in Norwegian or English

Ages: 2 Years to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2029-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Total difficulties score of the Strengths and Difficulties Questionnaire (SDQ) | [Time Frame: The SDQ is completed by both kindergarten teacher and each parent twice a year with approximately 6 months intervals during the three last year of attendance of the child in kindergarten, continued by the parents during the first two years i
  The SDQ has five scales (scored 0-10); emotional problems, conduct problems, hyperactivity, peer problems and pro-social scale. The scales are combined (excluding the pro-social scale) into a 'total difficulties' score (0-40).

CONTACTS AND LOCATIONS:
Overall Officials: Ingvar Bjelland, PhD, Principal Investigator — Haukeland University Hospital; Randi-Luise Møgster, MD, Study Director — Haukeland University Hospital
Locations (3):
- Norway (3):
  - Haukeland University Hospital, Bergen
  - Eventus Barnehage AS, Bergen
  - Øygarden municipality, Straume

REFERENCES:
- [Derived] Bjelland I, Wergeland GJ, Gillberg C, Gjestad R, Visnjic-Jevtic A, Lisaeth VK, Miniscalco C, Tufta ALF, Vermeer IL, Sadownik AR, Wilson P, Posserud MB. PRO-DIALOG-the effect of a novel dialogue-based parent-teacher conference on mental health in kindergarten children: a cluster randomized controlled trial. Trials. 2025 Aug 21;26(1):299. doi: 10.1186/s13063-025-08980-x. PMID 40842037
- See also: Paper that describes the development of the intervention / method under study in PRO-DIALOG — http://www.frontiersin.org/journals/psychiatry/articles/10.3389/fpsyt.2022.696531/full